CLINICAL TRIAL: NCT04304768
Title: Immune Dysfunction in HIV+ Opioid Users
Brief Title: Opioid, HIV and Immune System
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Savita Pahwa, Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20200178
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Immune Defect
Keywords: Flu vaccine response and HIV
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- HIV positive opioid users (Experimental): Participants will continue their standard of care antiretroviral therapy (ART) and receive flu vaccination as part of the study
  Interventions: Biological: Fluzone Quadrivalent
- HIV positive non-opioid users (Experimental): Participants will continue their standard of care antiretroviral therapy (ART) and receive flu vaccination as part of the study
  Interventions: Biological: Fluzone Quadrivalent
- HIV negative opioid users (Experimental): Participants will receive flu vaccination as part of the study
  Interventions: Biological: Fluzone Quadrivalent
- HIV negative non-opioid users (Experimental): Participants will receive flu vaccination as part of the study
  Interventions: Biological: Fluzone Quadrivalent

INTERVENTIONS:
Biological: Fluzone Quadrivalent — 0.5 ml prefilled syringe administrated intramuscularly
  Other Names: Influenza vaccination

SUMMARY:
The purpose of this research is to evaluate blood samples from HIV infected and non-HIV infected people opioid and non opioid users to understand how opioid affect the immune responses (body defenses against infection) to the flu vaccine.

ELIGIBILITY:
Inclusion Criteria:

For Opioid (OP) users/non-users:

1. OP users - prescribed opioids for at least the past 90 days; or injecting opioids for at least 90 days
2. Opioid never-users in the past year

Additional criteria for OP users:

1. OP use for 90 days pre-flu vaccination
2. Continued OP use for 4 weeks post flu vaccination

For HIV positive participants:

1) HIV infection, as documented by any licensed ELISA kit and confirmed by Western blot at any time prior to study entry. Participants on ART as a result of prior HIV documented infection will not be required to provide proof of diagnosis of HIV infection.

Additional criteria for HIV positive participants:

1. On ART for at least 1 year with plasma pending viral load (VL) <200 copies/mL. Occasional viral blips up to 1000 copies/ml also acceptable provided the patients are on continuing treatment
2. CD4 count available in the prior 6 months and >200/mm3
3. Undetectable viral load (< 200 copies/mL)

For HIV negative participants:

1) Documented negative HIV test, either by any licensed ELISA or rapid tests within the past 6 months.

For all participants:

1. Individuals age 18-60 yrs .
2. No history of other immunodeficiency disorders
3. Not on steroid or other immunosuppressive/immunomodulators medications.
4. No active malignancies.
5. No contraindication to receive influenza vaccination (allergy to chicken eggs or to any other substance of the vaccine).
6. Agreeable to receive the influenza vaccination.
7. Agreeable to participate in study for a complete course of study full visits.
8. Able to provide informed consent.

Exclusion Criteria:

1. Contraindication to receive influenza vaccination (allergy to chicken eggs or to any other substance of the vaccine).
2. Non-adherence to ART for HIV+
3. Unable to provide informed consent.
4. Other comorbid conditions such as diabetes mellitus type 2 (DMT2)
5. Influenza vaccination already given during the current vaccination season.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-11-18 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the antibody response | Baseline, 4 weeks, 6 months
  Antibody response as measured by the serum vaccine antigen specific hemagglutination inhibition antibody levels.

SECONDARY OUTCOMES:
Immune activation levels | Baseline
  Activation of T and B cells from peripheral blood mononuclear cells assessed via flow cytometry.
Inflammation biomarker levels | Baseline
  Plasma levels of Interleukin (IL)-6, IL-8, IL-12, IL-17, IL-22, Tumor necrosis factor (TNF) and monocyte activation markers soluble CD14 and soluble CD163 will be assessed via Magpix. All the biomarkers will be measured in nanograms/milliliter.
Circulating T follicular helper cell function | Week 4
  T follicular helper cell function measured from peripheral blood mononuclear cells via flow cytometry.
Circulating T follicular helper cell frequency | Week 4
  T follicular helper cell frequency measured from peripheral blood mononuclear cells via flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Savita Pahwa, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No